CLINICAL TRIAL: NCT01397994
Title: A Comparative Study to Assess the Efficacy of Nicorandil+Atenolol vs Atenolol in Treatment naïve Patients of Chronic Stable Angina.
Brief Title: Study to Assess Efficacy of Nicorandil+Atenolol vs Atenolol in Treatment of Chronic Stable Angina.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ferozsons Laboratories Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Tariq Ashraf, Assistant Professor Of cardiology, National Institute of Cardiovascular Diseases, Ferozsons Laboratories Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FZS NICORIL STUDY 01
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Stable Angina
Keywords: Nicorandil therapy in patients of chronic stable angina
MeSH Terms: conditions — Angina, Stable | interventions — Nicorandil; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicorandil test arm (Active Comparator): Nicorandil is given with atenolol therapy.
  Interventions: Drug: Nicorandil
- Atenolol control arm (Active Comparator): Atenolol 50 mg OD is given.
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Nicorandil — Patients would be advised 10mg bd nicorandil for the first seven days. Drug will be titrated to 20 mg bd after one week, atenolol 50 mg will be given along with nicorandil from day 1
  Other Names: Nicorandil/ Nicoril
  Arms: Nicorandil test arm
Drug: Atenolol — Patients in the control arm would be advised atenolol 50 mg od
  Other Names: Atenolol/Atenorm
  Arms: Atenolol control arm

SUMMARY:
This study is to determine the anti-anginal and anti-ischemic effect of k-channel opener, nicorandil in patients of chronic stable angina.

DETAILED DESCRIPTION:
Stress myocardial perfusion imaging (MPI) is widely used for the diagnosis and risk assessment of patients with known or suspected coronary artery disease (CAD). Also, MPI lends itself to monitoring the effects of therapeutic interventions such as anti-ischemic medications, gene therapy, and various percutaneous and surgical revascularization modalities.

The effects of nitrates, potassium channel activators, calcium-channel blockers, and beta-blockers on myocardial perfusion imaging are likely attributable to changes in myocardial blood flow and myocardial oxygen supply-demand ratio. The major anti-ischemic effect of BBs is a reduction in myocardial oxygen consumption both at rest and during stress. Beta-blockers decrease myocardial oxygen demand through a reduction in heart rate, blood pressure, and myocardial contractility. They also prolong diastole, therefore increasing coronary perfusion time. The effect of chronic atenolol use on dipyridamole SPECT MPI was assessed in a randomized, double-blind, crossover study that showed no difference in the perfusion defect size and severity between placebo and atenolol for the group as a whole, although one-third of patients had larger defects on atenolol than placebo. Bridges et al., 1992 (56)

Nicorandil, a potassium channel activator, when given for 3 weeks exhibited significant improvement in myocardial perfusion in both MI and angina patients, on exercise thallium scan. Yamazaki et al., 1993 (69).

Atenolol as shown in the cross over study does not affect myocardial perfusion significantly and hence combination therapy with nicorandil will help us to determine a significant benefit of nicorandil on MP. Results will be analyzed from base line in the same arm and the difference will be further compared with control arm.

Guidelines suggest beta blockers as first line of therapy. To assess the anti ischemic effects of nicorandil, combination therapy with atenolol will be compared with atenolol alone. Since atenolol effect on MP is insignificant an added advantage of nicorandil can be evaluated in comparative study.

Primary objective is to assess the anti ischemic effect of nicorandil.

The primary endpoint is to compare the anti ischemic effect over 4 weeks period.

Changes in perfusion will be evaluated in each arm at week 4 and comparison between the two study arms will be made to document the anti ischemic effects of nicorandil.

Primary efficacy variables of the study are the difference of the following endpoints from the baseline at week 4 and comparison between control and study arm using Ex- SPECT MPI.

Secondary efficacy variables of the study are the difference of the following endpoints from the baseline and comparison between control and study arm using ETT Bruce Protocol at week 4.

Secondary objectives of the study are to evaluate the anti anginal effect and safety of Nicorandil.

This is an open label, randomized controlled pilot study. Sponsor of this study is Ferozsons Labs. Ltd. All participating patients must sign a written informed consent form.

Eligible patients with proven CAD having at least one reversible or partially reversible myocardial perfusion defects on MPI SPECT - Tc-99m and functional class I & II of CSA, and laboratory values within predefined safety limits will be recruited.

Chief exclusion criteria include presence of only fixed perfusion defects, CSA functional class III and IV and prior revascularization.

A total of 40 patients will be enrolled in the study, 20 patients in each arm). Patients will be randomized in a 1:1 fashion to receive beta blocker in combination with nicorandil (experiment arm) or beta blocker (control arm) for four weeks until unacceptable toxicity, withdrawal of consent, whichever comes first.

Nicorandil dose will be titrated from 10mg bd for 7days to 20mg bd for next 3 weeks. Concurrent therapy for angina attacks will be allowed to be used with study medication.

All patients will have treadmill exercise using Bruce protocol. At peak exercise, 10-15 mCi of technetium - 99m tetrofosmin is injected and patient will exercise an additional 1 to 2 minutes.. Stress SPECT images will be acquired beginning 15 to 45 minutes after the completion of treadmill stress. At rest 30 mCi of technetium-99m tetrofosmin will be injected and SPECT images will be acquired using same protocol.

Study monitoring at the centre will be provided by the sponsor

ELIGIBILITY:
Inclusion Criteria:

1. Patients of chronic stable angina with abnormal Exercise Myocardial Perfusion Spect Scan with reversible and partially reversible ischemic changes.
2. Male and female
3. Age 25 to 65 years
4. Patient must understand and be willing, able and likely to comply with all study procedures and restrictions and comprehends the diary cards.
5. Patient must be able to give voluntary written informed consent.

Exclusion Criteria:

1. Hypertension of > 170/100 mm of Hg
2. Valvular heart disease and cardiomyopathy
3. Myocardial infarction in < 6 months
4. Unstable angina
5. Congestive cardiac failure
6. Severe anemia (Hb 7G/dl)
7. Cardiac arrhythmias or II or III degree AV block
8. Significant liver or renal dysfunction
9. IDDM (Type-1 diabetes mellitus)
10. Systolic blood pressure < 100 mm Hg
11. Pregnant and nursing women
12. Known hypersensitivity to nicorandil
13. On calcium channel blockers
14. Patients not eligible for Tc 99m SPECT
15. Patients in whom beta blockers are contraindicated
16. Geographical inaccessibility for treatment or follow-up evaluations

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
SPECT Tc99m- Tetrofosmin (MYOVIEW) | 4 weeks
  Changes in perfusion will be evaluated in each arm at week 4 and comparison between the two study arms will be made to document the anti ischemic effects of nicorandilusing Ex- SPECT MPI.
  * Improvement in SDS after 4 weeks of treatment (Summed Stress Score SSS, Summed Rest Score SRS, Summed Difference Score SDS)
  * Difference in number of reversible, partially reversible defects.
  * Improvement in the extent and severity of ischemic lesions.

SECONDARY OUTCOMES:
Exercise ECG Testing - Bruce protocol | 4weeks
  Secondary outcome measures of the study are the difference of the following endpoints from the baseline and comparison between control and study arm using ETT Bruce Protocol at week 4
  * Duration of exercise before the onset of angina or ST-segment depression (min)
  * Max. work load (Mets)
  * Max. ST depression (mm)
  * HR at max. ST depression (beats/min)
  * Syst. BP at max ST dep. (mm/Hg)
  other measures are:
  * Decrease in the frequency of anginal attacks
  * Use of rescue medicines
  * Adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Ashraf, MBBS,FCPS,FACC,FSCAI, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan